CLINICAL TRIAL: NCT05572957
Title: Left Bundle Branch Pacing as Initial Therapy in Patients With Non-ischemic Heart Failure and Left Bundle Branch Block (LIT-HF Study)
Brief Title: LBBP as Initial Therapy in Patients With Non-ischemic Heart Failure and LBBB
Acronym: LIT-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); West China Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Fujian Medical University Union Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstNanjingMU004
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Non-ischemic Cardiomyopathy; Heart Failure; Left Bundle-Branch Block
Keywords: Non-ischemic Cardiomyopathy; Heart Failure; Left Bundle-Branch Block; Guideline-Directed Medical Therapy; Left Bundle Branch Pacing; Implantable Cardioverter-Defibrillator; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDMT group (Active Comparator): With the current guidelines of recommended therapies for HF, each patient who meets the inclusion criteria should begin being on all 4 drug classes after enrollment, including a beta-blocker (BB), a RAS inhibitor (ACEI, ARB) or ARNI (preferred), an MRA, and an SGLT2i.
  The appeal drugs should be gradually uptitrated to the maximum tolerated dose within the first 3-6 months.
  Ivabradine will be added to the patients whose resting heart rates remain above 70 beats per minute (bpm) after adequate medical treatment, including a BB at maximum tolerated dose.
  Interventions: Drug: Guideline-Directed Medical Therapy(GDMT)
- LBBP+GDMT group (Experimental): In this arm, medications are the same as the GDMT group. The LBBP lead is introduced into the right ventricle (RV) and is placed on the right side of the interventricular septum (IVS). The lead is advanced deeply into the IVS until reaching the LV septal subendocardium and right bundle branch block (RBBB) morphology of the paced QRS complex is observed in electrocardiogram (ECG) lead V1.
  If LBBP fails, his bundle pacing (HBP) should be considered when HBP could correct LBBB.
  If both of LBBP and HBP fail, conventional BiVP-CRT could be the last option.
  Interventions: Combination Product: left bundle branch pacing combined with Guideline-Directed Medical Therapy(LBBP+GDMT)

INTERVENTIONS:
Drug: Guideline-Directed Medical Therapy(GDMT) — Quadruple anti-heart failure drug therapy: BB, ACEI/ARB/ARNI, MRA, and SGLT2i. If the initial dose according to guidelines is tolerated, the protocol would then direct the uptitration of medication dose over time to a specified target dose, unless not well tolerated.
  *Criteria for <3 months of optimized (complete) GDMT: 1) according to the latest management of HF, any of the "new quadruple therapy" is not used if the condition allowed; Or 2) the dose of any drug dose not reach the maximum tolerated target; Or 3) under the maximum tolerated dose of BB, ivabradine is not added with a heart rate still ≥70 bpm at rest.
  Other Names: Optimal Medical Therapy(OMT)
  Arms: GDMT group
Combination Product: left bundle branch pacing combined with Guideline-Directed Medical Therapy(LBBP+GDMT) — GDMT is the same as Drug intervention. LBBP is confirmed when: 1) the LBBB morphology disappeared and the paced RBBB pattern (typical or atypical) is observed in V1; and 2) LVAT is ≤100 ms at low output(≤3 V/0.5 ms); and at least 1 of the following is achieved: a) abrupt shortening of LVAT by >10 ms during mid/deep septal lead placement with a RBBB pattern in V1 at high output, which then remains short and constant at high and low output with further advancement of the lead to the final position; b) transition from nonselective to selective LBBP (QRS morphology transition from atypical RBBB to typical rsR' pattern in V1 and wide/large S-wave in V6 , with the appearance of an isoelectric segment and no LVAT change at high and low outputs); and c) transition from nonselective LBBP to LV septal pacing (lengthening of LVAT by at least 10 ms with or without obvious QRS morphology transition during threshold testing).
  HBP or BiVP is attempted using the standard-of-care technique.
  Arms: LBBP+GDMT group

SUMMARY:
The present study will recruit 50 symptomatic non-ischemic cardiomyopathy (NICM) patients with left ventricular ejection fraction (LVEF) below 35% and complete left bundle branch block (CLBBB), who have not received complete guideline-directed medical therapy (GDMT). Each patient was randomized to 2 groups, GDMT or left bundle branch pacing combined with GDMT (LBBP+GDMT) as initial therapy and was followed up for 2 phases: 0-6 months (phase I), 7-18 months (phase II). The primary objective is to compare the LVEF change , syncope and malignant ventricular arrhythmias between GDMT group and LBBP+GDMT group, and to observe which strategy will significantly reduce the percentage of recommendations for an implantable cardioverter-defibrillator (ICD) during phase I study. The second outcome measures including health economics, echocardiography parameters[left ventricular ejection fraction (LVEF), left ventricular end-systolic volume (LVESV), left ventricular end-diastolic volume (LVEDV)], N-terminal pro B-type natriuretic peptide (NT-proBNP) level, New York Heart Association (NYHA) class, 6-minute walking distance (6MWD), quality of life score(QOL) and incidence of clinical adverse events.

DETAILED DESCRIPTION:
Therapies currently approved to treat heart failure with reduced ejection fraction (HFrEF) have generally shown significant benefit on morbidity and mortality, resulting in strong recommendations in treatment guidelines. Four standard drugs classes, composed of beta-blockers, angiotensin-converting enzyme-inhibitor/angiotensin receptor blocker/angiotensin receptor-neprilysin inhibitor (ACE-I/ARB/ARNI), mineralocorticoid receptor antagonist (MRA) and sodium-glucose co-transporter 2 inhibitor (SGLT2i), have already been standard background therapy in HFrEF. Cardiac resynchronization therapy with pacemaker/Cardiac resynchronization therapy with defibrillation (CRT-P/CRT-D) is an established treatment to HF patients, especially in LVEF ≤35%, sinus rhythm, CLBBB with a QRS duration (QRSd) ≥150 ms, and symptoms on 3-6 months of GDMT. Both the 2021 ESC and the 2022 AHA/ACC/HFSA guidelines for HF included LVEF≤35% after 3-6 months of GDMT as a strong indication for ICD implantation in non-ischemic heart disease.

The traditional biventricular pacing (BiVP) could correct the cardiac dyssynchrony to improve clinical symptoms and reduce all-cause mortality in HF. However, almost 30%-40% of patients with successful implantation show no response and BiVP just corrects the mechanical dyssynchrony caused by LBBB not corrects the LBBB. His Purkinje conduction system pacing (HPCSP) technology has made significant progress in recent five years. His bundle pacing (HBP) and left bundle branch pacing(LBBP) can correct LBBB and achieve physiological cardiac resynchronization only by ordinary single-chamber or dual-chamber pacemaker. LBBP has been reported to produce stable pacing thresholds, adequately sensed R-wave amplitude, and higher likelihood to correct LBBB by pacing more distal to the site of conduction block compared with HBP. The feasibility and efficacy of LBBP for CRT in HF patients with LBBB was demonstrated by previous observational studies showing that LBBP-CRT achieves a narrower QRSd, higher percentage of super responders, and lower pacing thresholds than BiVP-CRT. The LBBP-RESYNC study showed that LBBP-CRT demonstrated greater LVEF improvement than BiVP-CRT in HF patients with NICM and LBBB.

It remains unclear as to the following questions: 1. After 3-6 months of GDMT, what is the percentage of patients with LVEFs improvement from ≤35% to >35% in HFrEF patients with NICM and CLBBB, and what are the absolute values of the increase in LVEFs; 2. How is the long-term prognosis of those patients with LVEF increased to >35% after GDMT. Whether these patients still need an ICD/CRT-D since they do not fall within the recommendations for primary prevention of sudden cardiac death (SCD); 3. What are the differences of LVEFs changes if LBBP is added to the medical treatment at the beginning.

There are to date no randomized studies comparing GDMT and LBBP combined with GDMT (LBBP+GDMT) as the initial therapy in HFrEF patients with NICM and CLBBB. The purpose of this study is to compare the therapeutic effects of LBBP+GDMT and GDMT on LV function and clinical endpoints in such patients. The present study will randomize about 50 patients in multiple centres to LBBP+GDMT group or GDMT group.

The study is divided into two phases:

Phase I (0-6 months) : Patients are randomly assigned to either the drug therapy group (GDMT group) or the experimental group (LBBP+GDMT group). In GDMT group at 3-month follow-up, CRT-P/CRT-D will be implanted if LVEF is still ≤35% with absolute increase <5% from baseline or ventricular tachycardia/ventricular fibrillation (VT/VF) events are recorded; otherwise, GDMT will be continued when LVEF >35% or LVEF≤35% but absolute increase >5% from baseline and no VT/VF event is observed. Patients in LBBP+GDMT group are directly treated with LBBP and GDMT after enrollment. The proportions of patients with LVEF ≤35% or VT/VF events in LBBP+GDMT group are assessed at 3-month and 6-month. The percentages of patients with LVEF ≤35% or VT/VF events in GDMT group are also assessed after 3 and 6 months as well.

Phase II (7-18 months): Patients in each group are followed up regularly (every 3-6 months, with mandatory at 12 and 18 months, with additional as appropriate) to assess the need for CRT-P/CRT-D/ICD when EF decreasing to ≤35%, syncope, or VT/VF events occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Non-ischemic cardiomyopathy with LVEF≤35% as assessed by echocardiography, NYHA class II-III, and less than 3 months of optimized (complete) GDMT*;
2. Sinus rhythm (paroxysmal atrial fibrillation may be present) with complete left bundle branch block meeting STRAUSS's criteria;
3. Between the ages of 18 and 80;
4. With informed consent signed.

Exclusion Criteria:

1. After mechanical tricuspid valve replacement;
2. Ischemic cardiomyopathy;
3. Persistent AF without AV node ablation;
4. History of unexplained syncope or indications for pacemaker implantation;
5. Indications for ICD implantation such as a history of sustained ventricular tachycardia or sudden cardiac arrest;
6. Unstable angina, acute MI, CABG or PCI within the past 3 months;
7. Enrollment in any other study；
8. A life expectancy of less than 12 months;
9. Pregnant or with child-bearing potential;
10. History of heart transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring ICD implantation for prevention of sudden cardiac death(SCD) | 6-month follow-up
  After treatment with two strategies(GDMT, LBBP+GDMT), the percentages of LVEF still ≤35% and/or ventricular arrhythmia events was assessed in both groups. That is, the percentage of patients who are eligible for primary/secondary prevention ICD implantation.

SECONDARY OUTCOMES:
Health economics | 3-month, 6-month, 12-month, and 18-month follow-up
  The cost of the two treatment strategies were evaluated comprehensively, including each inpatient, outpatient and unplanned follow-up
Changes in LVEF | Baseline; 3-month, 6-month, 12-month, and 18-month follow-up
  LVEF is assessed by echocardiography (Simpson's rule) and compared between the baseline and follow-up.
Changes in LVESV | Baseline; 3-month, 6-month, 12-month, and 18-month follow-up
  LVESV is assessed by echocardiography (Simpson's rule) and compared between the baseline and follow-up.
Changes in LVEDV | Baseline; 3-month, 6-month, 12-month, and 18-month follow-up
  LVEDV is assessed by echocardiography (Simpson's rule) and compared between the baseline and follow-up.
Changes in concentration of NT-proBNP in blood between baseline and follow-up | Baseline; 3-month, 6-month, 12-month, and 18-month follow-up
  Blood test is performed at each time frame to determine the concentration of NT-proBNP(unit: pg/mL)
Changes in New York Heart Association Heart Function Classification between baseline and follow-up | Baseline; 3-month, 6-month, 12-month, and 18-month follow-up
  The higher the classification, the more severe the heart failure symptoms(four levels: I, II, III and IV)
Change in Quality Of Life Questionnaire score between baseline and follow-up | Baseline; 3-month, 6-month, 12-month, and 18-month follow-up
  Reflect the effect of heart failure on quality of life, and higher scores represent a worse outcome
Incidence of clinical adverse events | Baseline; 3-month, 6-month, 12-month, and 18-month follow-up
  Including date and number of all-cause mortality, heart failure hospitalization, cardiovascular hospitalization and malignant ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Zou, MD,Ph.D, Principal Investigator — First Affiliated Hospital, Nanjing Medical University; Xiaofeng Hou, MD, Principal Investigator — First Affiliated Hospital, Nanjing Medical University; Yunlong Xia, MD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Yingxue Dong, MD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (6):
- China (6):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA. A Novel Pacing Strategy With Low and Stable Output: Pacing the Left Bundle Branch Immediately Beyond the Conduction Block. Can J Cardiol. 2017 Dec;33(12):1736.e1-1736.e3. doi: 10.1016/j.cjca.2017.09.013. Epub 2017 Sep 22. PMID 29173611
- [Background] Wang Y, Zhu H, Hou X, Wang Z, Zou F, Qian Z, Wei Y, Wang X, Zhang L, Li X, Liu Z, Xue S, Qin C, Zeng J, Li H, Wu H, Ma H, Ellenbogen KA, Gold MR, Fan X, Zou J; LBBP-RESYNC Investigators. Randomized Trial of Left Bundle Branch vs Biventricular Pacing for Cardiac Resynchronization Therapy. J Am Coll Cardiol. 2022 Sep 27;80(13):1205-1216. doi: 10.1016/j.jacc.2022.07.019. PMID 36137670
- [Background] Upadhyay GA, Vijayaraman P, Nayak HM, Verma N, Dandamudi G, Sharma PS, Saleem M, Mandrola J, Genovese D, Oren JW, Subzposh FA, Aziz Z, Beaser A, Shatz D, Besser S, Lang RM, Trohman RG, Knight BP, Tung R; His-SYNC Investigators. On-treatment comparison between corrective His bundle pacing and biventricular pacing for cardiac resynchronization: A secondary analysis of the His-SYNC Pilot Trial. Heart Rhythm. 2019 Dec;16(12):1797-1807. doi: 10.1016/j.hrthm.2019.05.009. Epub 2019 May 13. PMID 31096064
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499